CLINICAL TRIAL: NCT05868616
Title: Non-Invasive Method for Evaluation of Cardiac Resynchronization Therapy
Acronym: NIME-CRT
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); Norwegian Health Association (Other)
Responsible Party: Principal Investigator, Espen Remme, Dr.ing, Oslo University Hospital
Other Study IDs: 218564
Record Dates: First submitted 2023-04-26; First posted 2023-05-22 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure; Pacemaker DDD; Cardiomyopathies; Heart Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Heart Diseases; Cardiovascular Diseases | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Group 1 - Implantation: Patients admitted for CRT implantation according to current ESC/AHA guidelines
  Interventions: Device: Cardiac Resynchronization Therapy (CRT)
- Group 2 - 6 months control: Patients admitted for 6 months routine checkups of their CRT devices
  Interventions: Device: Cardiac Resynchronization Therapy (CRT)

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy (CRT) — Cardiac resynchronization therapy (CRT) is a modality of cardiac pacing used in patients with left ventricular (LV) systolic dysfunction and dyssynchronous ventricular activation that provides simultaneous or nearly simultaneous electrical activation of the LV and right ventricle (RV) via stimulation of the LV and RV (biventricular pacing) or LV alone.

SUMMARY:
Left bundle branch block (LBBB) exists in about 25% of patients with congestive heart failure and is associated with worsened prognosis. Cardiac resynchronization therapy (CRT) has been one of the most important advancements in the past two decades for patients with LBBB heart failure. However, 30-40% of patients receiving a CRT do not benefit from it. In this study, the investigators will test a noninvasive device to evaluate acute effect of CRT during implantation and at follow-up CRT controls. In addition, echocardiography will be performed during CRT turned ON and OFF to visualize the changes in intraventricular flow and functional parameters of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for CRT implantation or postoperative control at Oslo University Hospital based on the European Society of Cardiology (ESC) guidelines (2021), and criteria below:

  1. Sinus rhythm.
  2. New York Heart Association class II / III heart failure on diagnosis and on optimal medical therapy.
  3. Left bundle branch block.
  4. QRS duration ≥ 130 ms.
  5. Left ventricular ejection fraction ≤ 40%.
  6. Patients must have echocardiography examination before implantation
  7. Informed consent obtained from the patient.

Exclusion Criteria:

1. Age < 18 years and > 80 years;
2. Ongoing atrial fibrillation;
3. Complete atrioventricular block

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for CRT implantation according to European Society of Cardiology (ESC) guidelines (2021) or postoperative control at Oslo University Hospital.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Reverse remodelling at 6 months follow-up | 6 months
  Measured by left ventricular end-systolic volume reduction of at least 15% assessed by echocardiography

SECONDARY OUTCOMES:
Hospitalization | 2 years
  * all cause hospitalization
  * heart failure hospitalization defined by symptom, signs and biochemistry (NT-proBNP)
Mortality | 2 years
  * all cause death
  * sudden cardiac death
  * cardiovascular death
  * transplantation
New York Heart Association (NYHA) Functional Classification | 2 years
  The New York Heart Association (NYHA) functional classification provides a simple way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina.
Minnesota Living with Heart Failure Questionnaire | 2 years
  Minnesota living with heart failure questionnaire is a validated patient-oriented measure of the adverse effects of heart failure on a patient's life.
Packer clinical composite score | 2 years
  The Packer clinical composite score classifies each patient into 1 of 3 categories (improved, worsened, unchanged), and is determined using clinical outcomes (hospitalizations, death, heart transplant), heart failure status, and patient symptoms (defined by a higher New York Heart Association (NYHA) functional classification and quality of life measured using the Minnesota Living With Heart Failure Questionnaire). Each endpoint will be assessed at 6, 12, 18, and 24 months.
6 minute walk test | 6 months
  The 6 minute walk test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. The test will be performed in group 1 before implantation and at 6 months control to evaluate response to intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Espen W. Remme, Dr.ing, Study Director — Oslo University Hospital; Marit Witso, MD, Principal Investigator — Oslo University Hospital; Hongxing Luo, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT05868616/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT05868616/ICF_001.pdf